CLINICAL TRIAL: NCT00118807
Title: Randomized Trial of the Effectiveness of Amodiaquine-Artesunate, Amodiaquine-Sulfadoxine-Pyrimethamine, and Chloroquine-Sulfadoxine-Pyrimethamine, for Treatment of Uncomplicated Malaria in Gambian Children
Brief Title: Trial of the Effectiveness of AQ/AS, SP/AQ and SP/CQ for Uncomplicated Malaria in Gambian Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); National Malaria Control Programme, The Gambia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC940; MRC SCC No. 940
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2003-06

CONDITIONS: Malaria
Keywords: malaria treatment; artemisinin based combination therapy; Plasmodium falciparum; pragmatic trial; effectiveness
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Amodiaquine; Artesunate; fanasil, pyrimethamine drug combination; Chloroquine

INTERVENTIONS:
Drug: Amodiaquine plus artesunate (AQ/AS)
Drug: Sulfadoxine-pyrimethamine plus chloroquine (SP/CQ)
Drug: Sulfadoxine-pyrimethamine plus amodiaquine (SP/AQ)

SUMMARY:
The purpose of this trial is to compare the effectiveness of three combination treatments for uncomplicated malaria when given in operational settings, without supervision of doses other than the first dose.

DETAILED DESCRIPTION:
Children aged 0.5-10 years presenting at health centres with fever or history of fever and other symptoms suggestive of malaria will be screened; children found to have uncomplicated Plasmodium falciparum malaria will be randomized to receive treatment with AS/AQ, SP/AQ or SP/CQ. A drug dispenser will supervise the first dose of medication and subsequent doses will be given to the child's parent to be administered at home, unsupervised by the study team. Patients will be visited at home three days later. Unused medication will be counted and the mother will be asked about the number of doses the child received and any side effects. Children will be seen again 2 and 4 weeks after treatment to collect finger prick samples for packed cell volume (PCV) and malaria microscopy. The primary endpoint is clinical failure by day 28. Analysis will be by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Presentation at health centre with febrile illness
* Monoinfection with P. falciparum
* Parasitaemia >=500/microlitre
* Fever or history of fever

Exclusion Criteria:

* Signs of severe or complicated malaria (persistent vomiting with or without dehydration, history of convulsion during the present illness, inability to sit or stand, parasitaemia >200,000/ul)
* Severe malnutrition
* Clinically evident concomitant disease
* PCV <20%
* History of allergy to the study medications
* Residence outside the study area and hence difficult to follow up

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1800
Dates: Start 2003-08; Study Completion 2004-02

PRIMARY OUTCOMES:
Clinical failure by day 28
Incidence of adverse events

SECONDARY OUTCOMES:
Compliance with treatment regimen
Parasitological failure by day 28
Clinical failure by day 14
Parasitological failure rate by day 14
Mean PCV on day 28
Gametocyte carriage rates
Transmissibility after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sam K Dunyo, PhD, Principal Investigator — Medical Research Council; Paul J Milligan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Medical Research Council Laboratories, Banjul, City of Banjul, The Gambia